CLINICAL TRIAL: NCT00542971
Title: Phase I-II Study of Idarubicin, Cytarabine, and Sorafenib (BAY43-9006), an Oral Vascular Endothelial Growth Factor (VEGF), Rapidly Accelerated Fibrosarcoma (RAF) and FMS-like Tyrosine Kinase 3 (FLT3), in Patients With High-risk MDS and AML
Brief Title: Phase I-II Study of Idarubicin, Cytarabine, and Sorafenib (BAY43-9006)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0977
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: AML; Acute Myeloid Leukemia; Myelodysplastic Disorders
Keywords: Leukemia; AML; High-Risk MDS; Acute Myeloid Leukemia; High-Risk Myelodysplastic Disorder; Idarubicin; Ara-C; Cytarabine; Sorafenib; BAY43-9006
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Idarubicin; Sorafenib; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + Idarubicin + Ara-C (Experimental): Sorafenib starting dose 400 mg orally for 7 days; Idarubicin 12 mg/m^2 intravenous (IV) daily (days 1-3); and Ara-C 1.5 g/m^2 IV over 24 hours daily (days 1-4)
  Interventions: Drug: Idarubicin; Drug: Sorafenib; Drug: Ara-C

INTERVENTIONS:
Drug: Idarubicin — 12 mg/m^2 IV over 1 hour daily (days 1-3)
  Other Names: Idamycin®
Drug: Sorafenib — Starting dose 400 mg by mouth for 7 days
  Other Names: Nexavar®
Drug: Ara-C — 1.5 g/m^2 IV over 24 hours daily (days 1-4)
  Other Names: Cytarabine; Cytosar-U®; Arabinosylcytosine

SUMMARY:
A primary goal of this clinical research study is to find the highest safe dose of sorafenib that can be given in combination with idarubicin and Ara-C for the treatment of acute myelogenous leukemia (AML) and high-risk, myelodysplastic syndrome (MDS).

Once the highest safe dose is found, researchers will then try to learn if this combination treatment can help control AML and high-risk MDS in newly diagnosed patients. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Sorafenib is designed to block the function of important proteins in cancer cells. When active, these proteins help cause abnormal growth and behavior of leukemia cells.

Idarubicin and Ara-C are both designed to insert themselves into DNA (the genetic material of cells) and to stop DNA from repairing itself.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study.

If you are enrolled in the Phase I part of this study, the dose of sorafenib you receive with Ara-C and idarubicin will depend on when you enrolled in this study. Each new group of 3 participants will receive a higher dose level of sorafenib than the previous group until the highest safe dose of sorafenib that can be given in combination with Ara-C and idarubicin is reached.

If you are enrolled in the Phase II portion of this study, you will receive the highest safe dose of sorafenib in combination with Ara-C and idarubicin found in the Phase I part.

Study Drug Administration:

During the study, you will receive treatment over 28-day "cycles." The doses of idarubicin and Ara-C are the same for all study participants.

On Days 1-4 (Days 1-3 if you are older than 60) of each induction cycle (#1 and possibly #2), you will receive Ara-C through a nonstop infusion (through a needle in your vein). You will also receive steroids by mouth or through a vein every day to reduce the risks of side effects, such as rash.

On Days 1-3 of each induction cycle (#1 and possibly #2), you will receive idarubicin by vein over 1 hour once a day.

In general, sorafenib will be taken by mouth twice daily on Days 1-7, unless otherwise instructed. However, the dose of sorafenib may differ among study participants. Sorafenib should be taken with water on an empty stomach. Your study doctor will give you complete instructions on when and how to take sorafenib.

Depending on the side effects that you may have, the dose of sorafenib may be decreased, stopped until side effects go away, or even stopped completely, if your doctor thinks that this is in your best interest.

Study Visits:

During Cycles 1-2, you will have study visits about 2 times a week. You may need to have study visits more often when the study doctor thinks it is necessary. At these visits, you will have the following procedures performed.

* You will be asked about any side effects you may have experienced and any medications you may be taking.
* Blood (about 2 teaspoons) will be drawn for routine tests.

During Cycles 1 and 2, between Days 21-28, you will have a bone marrow aspirate and/or biopsy performed to check the status of the disease.

For Cycle 3 and in further cycles, you will have a bone marrow aspirate as determined necessary by your doctor. If your doctor thinks you have responded to the treatment, you will then have bone marrow aspirates collected every 3-6 months, if your doctor feels this to be necessary.

Consolidation Therapy:

If it is found that the disease is responding to treatment, you may receive 5 additional cycles of therapy. These cycles are called "consolidation" therapy and will be given every 4-6 weeks.

On Days 1-3, Ara-C will be given as a nonstop infusion. You will also receive steroids either by mouth or by vein to help reduce the risk of side effects.

On Days 1-2, idarubicin will be given by vein over 1 hour.

Sorafenib will be taken twice daily by mouth for 7 or more days, at a schedule determined by your study doctor.

After each cycle, about every 4-6 weeks, blood (about 2 teaspoons) will be drawn to check your blood count levels.

Maintenance Therapy:

After 5 cycles of consolidation therapy, and according to your response to consolidation therapy, you may continue on this study to receive "maintenance" treatment, as needed, and as determined by your study doctor for up to 7 more cycles.

You will take sorafenib twice a day every day during the 28-day cycle.

Every 1-4 weeks, blood (about 2 teaspoons) will be drawn for routine tests.

Length of Study:

You may receive up to 14 cycles in total of therapy. You may be taken off this study if the leukemia gets worse, develop another illness that interferes with taking the study drugs, or you have intolerable side effects.

This is an investigational study. Sorafenib is FDA approved and commercially available for the treatment of metastatic renal cancer only. Idarubicin is FDA approved for use in combination with other approved antileukemic drugs for the treatment of acute myeloid leukemia (AML) in adults. Cytarabine is FDA approved for use in the treatment of leukemia. The use of sorafenib combined with idarubicin and Ara-C in the treatment of AML and high-risk MDS is investigational and authorized for use in research only. Up to 75 patients will take part in this study. All patients will be enrolled at M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of 1) AML (World Health Organization classification definition of > 20% blasts), or 2) high risk MDS (defined as the presence of > 10% blasts).
2. Patients aged 15 to 60 years are eligible. Patients older than 60 who are deemed fit to receive intensive chemotherapy by the treating physician are eligible after discussion with the Principal Investigator (PI). For the Phase II portion of the study, patients must be chemo-naïve, i.e. not have received any prior chemotherapy (except hydrea) for AML or MDS. They could have received hypomethylator agents, transfusions, hematopoietic growth factors or vitamins. Temporary prior measures such as pheresis or hydrea are allowed. In the Phase I portion, patients with relapsed or refractory AML/MDS are also eligible.
3. Serum biochemical values with the following limits unless considered due to leukemia: 1) creatinine less than or equal to 2 mg/dl, 2) total bilirubin less than or equal to 2 mg/dL, unless increase is due to hemolysis or congenital disorder, and 3) transaminases (SG PT) less than or equal to 2.5 times upper limit of normal (ULN)
4. Ability to take oral medication.
5. Ability to understand and provide signed informed consent.
6. Baseline test of ejection fraction must be >/=50%.
7. Performance status < 3, unless directly related to the disease process as determined by the principal investigator.

Exclusion Criteria:

1. Patients with Acute promyelocytic leukemia (APL).
2. Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results.
3. Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, Intrauterine Device (IUD), diaphragm, abstinence, or condoms by their partner) over the entire course of the study.
4. Any significant, uncontrolled hypertension.
5. Cardiac disease: Congestive heart failure > class II The New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
6. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy. Sorafenib is contraindicated in patients with known severe hypersensitivity to sorafenib or any of the excipients.
7. Known human immunodeficiency virus (HIV) infection or active Hepatitis B or C.
8. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
9. Pulmonary hemorrhage/bleeding event > or = to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks of first dose of study drug.
10. Any other hemorrhage/bleeding event > or = to CTCAE Grade 3 within 4 weeks of first dose of study drug.
11. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
12. Use of St. John's Wort or rifampin.
13. Known or suspected allergy to sorafenib or any agent given in the course of this trial.
14. Active clinically serious and uncontrolled infection > CTCAE Grade 2
15. Serious non-healing wound, ulcer, or bone fracture

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2007 to February 2009. All participants were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 78 participants registered on this study, three (3) were excluded prior to receiving treatment.
Groups:
- Sorafenib + Idarubicin + Ara-C: Sorafenib starting dose 400 mg orally for 7 days; Idarubicin 12 mg/m2 intravenous (IV) daily (days 1-3); and Ara-C 1.5 g/m2 IV over 24 hours daily (days 1-4)
Period: Overall Study
Arm/Group | Sorafenib + Idarubicin + Ara-C
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib + Idarubicin + Ara-C
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 52 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is dose level where grade 3-4 sorafenib-attributable toxicity in <2 of 6 participants. Dose-Limiting Toxicity graded according to the NCI Common Toxicity Criteria version 3.0.
Time Frame: Twice a week for first two 28 day cycles
Population: 10 participants were treated with escalating doses of sorafenib with chemotherapy to establish the feasibility of the combination.
Measure: Number; unit: milligrams/twice a day (BID)
Arm/Group | Sorafenib + Idarubicin + Ara-C
Number analyzed (Participants) | 10
milligrams/twice a day (BID) | 400

2. Secondary Outcome: Number of Participants With Complete Response
Description: Complete response was defined by the presence of < 5% blasts in the bone marrow (BM) with > 1 x 10^9/L platelets in the peripheral blood (PB).
Time Frame: Baseline to 2 years or disease progression.
Measure: Number; unit: Participants
Arm/Group | Sorafenib + Idarubicin + Ara-C
Number analyzed (Participants) | 75
Participants
  Complete Response | 54
  No Complete Response | 21

ADVERSE EVENTS:
Time Frame: 2 years, 4 months.
Arm/Group | Sorafenib + Idarubicin + Ara-C
Serious Adverse Events (participants affected / at risk) | 8/78
Other Adverse Events (participants affected / at risk) | 47/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Idarubicin + Ara-C (N=78)
Infection (Infections and infestations) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Death (Gastrointestinal disorders) | 3 (3) — All events were unrelated to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Idarubicin + Ara-C (N=75)
Diarrhea (Gastrointestinal disorders) | 23 (26)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (4)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 27 (40)
Rash Hand Foot Reaction (Skin and subcutaneous tissue disorders) | 9 (11)
Cardiac General (Cardiac disorders) | 1 (1)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 2 (2)
Opportunistic Infection (Infections and infestations) | 12 (12)
Infection (Infections and infestations) | 8 (9)
Rash Desquamation (Skin and subcutaneous tissue disorders) | 15 (15)
Mucositis (Gastrointestinal disorders) | 7 (7)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 2 (2)
Elevated Creatinine (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage Bleeding (Blood and lymphatic system disorders) | 4 (4)
Bilirubin (Metabolism and nutrition disorders) | 6 (6)
edema (Blood and lymphatic system disorders) | 5 (5)
Mood Alteration (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 3 (3)
Death (General disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pain (General disorders) | 3 (7)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Tumor Lysis Syndrome (General disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 2 (2)
Dysphasia (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cardiac Ischemia/Infarct (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No